CLINICAL TRIAL: NCT04784741
Title: Effect of Low Amplitude Vibration Therapy on Flexibility of Hamstring Muscle in Athletes of Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Clinical Research Center (Other)
Responsible Party: Principal Investigator, Dr Jaweria Syed, Principal Investigator, Shifa Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/00255
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Hamstring Contractures; Whole Body Vibration
Keywords: whole body vibration; Hamstring flexibility; ROM; Balance; Postural stability index

STUDY DESIGN:
Intervention Model Description: A total of 40 were included in the study who full filled the inclusion criteria, athletes were randomly assigned into two groups: Control and Experimental group. Additionally, data was collected from healthy athletes doing their training at Pakistan Sports Board, Islamabad.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The control group was given the static hamstring muscle stretches, five sessions on alternative days according to the set protocols.
  Interventions: Other: Conventional static hamstring muscle stretching; Device: Biodex Balance System; Procedure: Range of motion of hamstring muscle
- Experimental Group (Experimental): Given five sessions of low amplitude whole body vibration therapy for duration of 10 minutes, on alternative days, along with static stretching of hamstring muscles.
  Interventions: Device: Low amplitude whole body vibration therapy; Device: Biodex Balance System; Procedure: Range of motion of hamstring muscle

INTERVENTIONS:
Other: Conventional static hamstring muscle stretching — Static stretching protocol had 10 repetitions in total with 15 seconds stretch time and 30 seconds relaxing time of hamstring muscle.
  Arms: Control group
Device: Low amplitude whole body vibration therapy — Given five sessions of low amplitude whole body vibration therapy for duration of 10 minutes, on alternative days, along with static stretching of hamstring muscles.
  Static stretching protocol had 10 repetitions in total with 15 seconds stretch time and 30 seconds relaxing time of hamstring muscle.
  Arms: Experimental Group
Device: Biodex Balance System — Pre and post balance assessment by Biodex balance system
Procedure: Range of motion of hamstring muscle — Straight Leg Raising to check pre and post Range of Motion by using Goniometer

SUMMARY:
Whole body vibration therapy is rapidly becoming a topic of interest for the researchers around the world. Evidence suggests that Whole body vibration has an effect on improving flexibility of hamstring muscle and balance in athletes. The purpose was to examine the effect of low amplitude Whole body vibration on the flexibility of hamstring muscle and improving balance in athletes of Pakistan

DETAILED DESCRIPTION:
A total 60 number of athletes were analyzed and out of these 40 were included in the study who full fill the inclusion criteria, selected athletes were randomly assigned into two groups (control & experimental). After a total 2 drop outs from control group and 3 drop outs from experimental group, there were 18 athletes in control group and 17 in experimental group who continued till the analysis. Experimental group was given five sessions of low amplitude whole body vibration therapy for almost duration of 10 minutes, on alternative days, along with static stretching of hamstring muscles for 5 minutes and the control group was given only the static hamstring muscle stretches for five minutes, and same five sessions alike on alternative days. Static stretching protocol had 10 stretches in total with 15 seconds stretch time and 30 seconds relaxing time of hamstring muscle. All participants were assessed using Biodex Whole body vibration plate, Biodex balance system , Goniometer and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* National athletes of Pakistan.
* Age between 18-30 years

Exclusion Criteria:

* Athletes having history of any acute injury within last 6 weeks.
* Athletes who have had any surgical procedure previously or Patients who were medically unstable.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Pre Range of Motion of hamstring muscle (ROM) | outcome at baseline (day zero)
  The outcome was the pre status of flexibility in hamstring muscle assessed using Goniometer.
Post Range of Motion of hamstring muscle (ROM) | outcome at the end of 10 days
  The outcome was the post status of flexibility in hamstring muscle assessed using Goniometer.
Pre Balance | outcome at baseline (day zero)
  The outcome was pre balance testing using biodex balance system.
Post Balance | outcome at the end of 10 days
  The outcome was post balance testing using biodex balance system.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaweria Syed, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR